CLINICAL TRIAL: NCT05956236
Title: Hip Prospective Study: Long-term Post-market Clinical Follow-up on the Use of SERF Hip Prostheses
Brief Title: Hip Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: HiPS
Record Dates: First submitted 2023-03-23; First posted 2023-07-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Hip Arthropathy
Keywords: Hip arthropalsty; Hip Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In an evaluation report dated 2014, the HAS (Haute Autorité de Santé -French National Authority for Health) highlights that long-term clinical data on hip prostheses are needed in the context of the French healthcare system. In addition, per the European Regulation 2017/745, medical devices manufacturers shall conduct Post-Market Clinical Follow-up (PMCF) on their devices or provide a justification why PMCF is not applicable.

Therefore, as part of the PMCF process of their hip prostheses, SERF wants to conduct a PMCF investigation to ensure the long-term real-life performance, safety and benefits of these prostheses.

HiPS is a non-comparative, prospective, multicentric, national, 15-year follow-up clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* Planned to be implanted with investigational medical devices per the IFUs:

  * Implantation in skeletally mature adults (usually aged 60-65 and over), with an extremely painful and/or disabled joint and insufficiently improved by alternative treatment options after an observation period lasting from a few weeks to a few months
  * Implantation of investigational medical devices as integrated systems (all components from SERF, no component from another manufacturer)
  * For an intended purpose and indication listed in the IFUs
* Affiliated to French social security
* Who provided a dated and signed informed consent form

Exclusion Criteria:

* Patient protected by a French legal measure
* Patient not able to express his/her consent as deemed by the investigator
* Patient deprived of liberty or hospitalized without consent
* Pregnant or breastfeeding women
* Patient contraindicated to investigational medical devices implantation per the IFUs
* Patient contraindicated to radiographic follow-up
* Patient a priori not able to meet the follow-up visits as deemed by the investigator
* Patient not able to fulfil a self-assessment questionnaire as deemed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients corresponding to the target treated population of the investigational medical devices, planned to be implanted with investigational medical devices per the Instructions for Use (IFU), who can participate to a clinical investigation, are not vulnerable and can meet the follow-up visits (a priori) and fulfil a self-assessment questionnaire will be included.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2046-04 (Estimated); Study Completion 2046-04 (Estimated)

PRIMARY OUTCOMES:
Survival rate | Per operative period to 15 years
  To assess the survival rate of the investigational medical devices at the end of their claimed implantation duration

SECONDARY OUTCOMES:
Intermediate survival rates | Per operative period to 10 years
  To assess the survival rate of the investigational medical devices at the intermediate timepoints
Functional improvement | Per operative period to 15 years
  To assess the evolution of patient's functional capacity post-implantation using HOOS score
Functional improvement | Per operative period to 15 years
  To assess the evolution of patient's functional capacity post-implantation using Harris Hips score
Functional improvement | Per operative period to 15 years
  To assess the evolution of patient's activity post-implantation using UCLA scale
Functional improvement | Per operative period to 15 years
  To assess the evolution of patient's activity post-implantation using Charnley score
Leg length discrepancy | Pre operative period to 15 years
  To assess patient's leg length discrepancy post-implantation (visual evaluation)
Patient's Pain | Pre operative period to 15 years
  To assess patient's pain (Visual Analogic Scale)
Patient's quality of life | Pre operative period to 15 years
  To assess patient's quality of life post-implantation (Forgotten Joint Score)
Patient's satisfaction | Post operative period to 15 years
  To assess patients' satisfaction with the operation (4-points question)
Surgeon's satisfaction | Per operative period to 15 years
  To assess surgeons' satisfaction with the operation
Adverse events | Per operative period to 15 years
  To assess the long-term safety of investigational medical devices as well as post-operative safety of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU St Etienne, Saint-Priest-en-Jarez, France